CLINICAL TRIAL: NCT07162467
Title: Tryptophan-Kynurenine Pathway Metabolism in the Pathophysiology of Cognitive Impairment in Schizophrenia.
Status: Enrolling by invitation | Type: Observational
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FESW-TKAH
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognitive funciton; tryptophan-kynurenine pathway
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Schizophrenic Patients: 100 eligible individuals will meet DSM-5 criteria for schizophrenia or schizoaffective disorder, be Han Chinese aged 18-55 years, presenting with a first episode of illness ≤ 5 years duration. Prior antipsychotic exposure must be ≤ 4 weeks cumulatively, or patients must be treatment-naïve. Informed consent will be obtained from patients and their families.
- Healthy Control: 100 healthy, age-, gender-, and education-matched Han Chinese volunteers, with informed consent.

SUMMARY:
Schizophrenia is a common, long-term mental illness. It causes problems with thoughts, feelings, and behavior, including positive symptoms (hallucinations, delusions), negative symptoms (lack of emotion, motivation), and cognitive impairment (trouble with thinking, memory, and attention). While antipsychotic drugs effectively treat positive symptoms, they don't help much with cognitive impairment.This study will examine how the tryptophan-kynurenine pathway in the brain contributes to cognitive problems in people having their first episode of schizophrenia and treated with a single antipsychotic. Our goal is to create models for early detection of cognitive impairment in schizophrenia and find potential targets for new treatments to improve thinking and memory.

DETAILED DESCRIPTION:
This single-center, prospective study will recruit 100 treatment-naïve, first-episode schizophrenia (SZ) patients at Tianjin Anding Hospital for an 8-week follow-up. All patients will receive monotherapy with risperidone and undergo baseline and week 8 assessments including clinical rating scales and the MATRICS Consensus Cognitive Battery (MCCB), along with peripheral blood sample collection. Concurrently, 100 age-, sex-, and education-matched healthy controls (HCs) will be recruited. Prior data from 300 medication-naïve SZ patients and 100 HCs will be selectively included in the final analysis (totaling 300 SZ patients and 200 HCs). We hypothesize that dysregulation of the tryptophan-kynurenine (TRP-KYN) pathway in SZ patients, leading to an imbalanced ratio of neuroprotective kynurenic acid (KYNA) to neurotoxic quinolinic acid (QUIN), affects inflammatory markers and NMDA receptor (NMDAR) levels, ultimately causing cognitive impairment. Specifically, we will analyze the association between cognitive function and plasma TRP-KYN pathway metabolites in medication-naïve FES patients; relationship between cognitive function and TRP-KYN pathway gene polymorphisms and mRNA expression in medication-naïve FES patients; and changes in cognitive function post-8-week treatment with plasma TRP-KYN pathway mRNA expression and metabolite levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers matched to the patient group on sex, age, and education level;
* Ethnic Han Chinese;
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Significant comorbid medical or neurological conditions;
* Any DSM-5-defined psychiatric disorder;
* Family history of psychiatric illness spanning three or more generations;
* Current use of psychoactive medications;
* Refusal to provide informed consent/participate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will recruit 100 Han Chinese adults aged 18-55 years for two cohorts: patients and healthy controls. The patient cohort will comprise individuals experiencing their first episode of schizophrenia or schizophreniform disorder with a duration of ≤ 5 years, who have either never received antipsychotic treatment or have received it for a cumulative duration of ≤ 4 weeks prior to enrollment. Recruitment will be conducted from the outpatient and inpatient services of Tianjin Anding Hospital and surrounding communities in Tianjin, China. The healthy control cohort will consist of 100 Han Chinese adults matched to the patient group for sex, age, and education. These individuals must have no personal or family history of major psychiatric disorders and demonstrate no cognitive impairment on formal testing.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
TRP-KYN pathway candidate plasma metabolite levels | Baseline, week8
  Plasma levels of tryptophan-kynurenine (TRP-KYN) pathway candidate metabolites, including kynurenine, kynurenic acid, kynurenic quinolinic acid, quinolinic acid, tryptophan, indole-3-acetic acid, and indole-3-propionic acid, were quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS). Sample information was registered in MetLIMS software, with designated positions for samples of interest, blanks, standards, and quality control samples. Samples were added to corresponding wells in a 96-well plate provided in the kit. Subsequently, derivatization was performed by adding a 5% phenylisothiocyanate solution. Finally, target analytes were extracted with an organic solvent and diluted. The pre-processed sample extracts underwent High-Performance Liquid Chromatography-Mass Spectrometry detection. Each sample was analyzed in two parts: the first involved signal acquisition in flow injection analysis mode, and the second in liquid chromatography-mass spectrometry mode.
Cognitive Function | Baseline, week8
  All participants underwent cognitive function assessment based on the MATRICS Consensus Cognitive Battery (MCCB). The MCCB is a standardized instrument for assessing cognitive function in schizophrenia. It comprises nine subtests primarily evaluating seven cognitive domains: processing speed, attention/alertness, working memory, verbal learning, visual memory, reasoning and problem-solving, and social cognition. The MCCB scoring procedure generates standardised T-scores that are corrected for age, gender, and educational level. Higher T-scores indicate better cognitive function.
Candidate gene mRNA expression levels | Baseline, week8
  Whole blood was collected in BD PAXgene® Blood RNA tubes (2.5 mL from antecubital veins) and gently inverted to mix. Samples were incubated vertically at room temperature for 2 hours, then stored at -20°C overnight before transfer to -80°C for RNA extraction. Extracted RNA was reverse transcribed to synthesize cDNA. Gene expression levels of TDO, IDO, KMO, KAT-II, KYNU, and 3HAO were determined by RT-qPCR with gel electrophoresis for product validation and densitometric scanning using a gel imaging system.

SECONDARY OUTCOMES:
Psychiatric Symptoms | Baseline, week8
  The psychiatric symptoms of schizophrenia were assessed in all enrolled patients using the Positive and Negative Syndrome Scale (PANSS). The PANSS is a 30-item clinician-rated scale yielding a total score ranging from 30 (least symptomatic) to 210 (symptomatic), where higher scores indicate more severe psychopathology.
Depressive Symptoms | Baseline, week8
  The Hamilton Depression Scale-24 (HAMD-24) was used to assess the severity of depressive symptoms. Each item was scored on a scale of 0 (none) to 4 (severe); the total score ranged from 0 to 76, with higher scores indicating more severe depressive symptoms.
Anxiety Symptoms | baseline, week 8
  The Hamilton Anxiety Scale (HAMA) is used to assess the severity of anxiety symptoms. Each item is scored on a scale of 0 (none) to 4 (very severe), with a total score range of 0-56. Higher scores indicate more severe anxiety symptoms.
Clinical Global Impression of Efficacy | baseline, week 8
  The Clinical Global Impression (CGI) scale is used to assess treatment outcomes in patients, particularly for monitoring efficacy in severe mental disorders such as schizophrenia. The CGI encompasses three core dimensions: Severity of Illness (SI), Global Improvement (GI), and an Efficacy Index (EI). The CGI provides a structured assessment framework for healthcare professionals through a quantitative scoring system. In particular, the CGI-EI integrates therapeutic effects with adverse events, resulting in a graded assessment ranging from 0 (Markedly worse) to 4 (Markedly improved), suitable for monitoring during the entire course of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, China